CLINICAL TRIAL: NCT06262074
Title: Effect of Structured Training Program on Functional Abilities in Patients With Diabetic Neuropathy
Brief Title: Effect of Structured Training Program in Diabetic Patients
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Maharishi Markendeswar University (Deemed to be University) (Other)
Responsible Party: Principal Investigator, Subhasish Chatterjee, Clinical Professor, Maharishi Markendeswar University (Deemed to be University)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IEC-2418
Record Dates: First submitted 2024-01-31; First posted 2024-02-15 (Actual); Last update posted 2024-02-15 (Actual); Status verified 2024-02

CONDITIONS: Diabetic Peripheral Neuropathy

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group-1 (Structured Exercise Program) (Experimental): Patients undergo structured exercise sessions lasting 30 minutes, encompassing activities such as range of motion, flexibility exercises, strength training, balance exercises, and aerobic exercises, with designated intervals between each session.
  Interventions: Other: Structured Exercise Program
- Group-2 (Non-Structured Exercise Program) (Other): Patients are provided with a simple exercise routine that lacks a structured format.
  Interventions: Other: Non structured exercise program

INTERVENTIONS:
Other: Structured Exercise Program — 30 minutes of structured exercise programs
  Arms: Group-1 (Structured Exercise Program)
Other: Non structured exercise program — Non structured exercises
  Arms: Group-2 (Non-Structured Exercise Program)

SUMMARY:
Diabetic neuropathy, a challenging condition resulting from poorly managed type-1 or type-2 diabetes mellitus, often proves resistant to conventional medications when it comes to alleviating the associated symptoms. In such cases, implementing a well-organized exercise regimen has proven beneficial in mitigating diverse symptoms associated with the condition and enhancing the overall quality of life for affected individuals.

DETAILED DESCRIPTION:
The goal of this type of interventional study is to assess the effect a well-defined exercise program for individuals with DPN, despite the existence of various individualized exercise programs designed for DPN patients. The main questions this study aims to answer is:

What is the effect of a 4-weeks structured training program as an adjunct to general lower limb exercise in patients with DPN on pain, sensory symptoms, balance, vibration sense and Quality of life?

Group 1:

Patients in group 1 will receive a structured exercise program.

Group 2:

Patients in group 2 will receive a non-structured exercise program. This group will allow us to compare the effects of a structured and a non-structured exercise program.

ELIGIBILITY:
Inclusion Criteria:

* Diabetes mellitus with moderate to severe DPN
* Subjects of both gender
* Age from 40 to 70 years
* Independent walking
* MNSI score more than 2 out of 13

Exclusion Criteria:

* Presence of an active planter ulcer
* History of surgery during intervention period
* Neurological diseases other than DPN

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-02-08 (Actual); Primary Completion 2024-02-08 (Actual); Study Completion 2024-03-31 (Estimated)

PRIMARY OUTCOMES:
Michigan neuropathy screening instrument (MNSI) | The measurement will be taken during the baseline assessment and again after the completion of treatment.
  The scale consists of two parts: the first part involves a patient history assessment, while the second part focuses on physical examination. This scale is considered both reliable and practical for evaluating the severity of neuropathy. If the patient's score increases, it indicates a higher severity of the disease, whereas if the score decreases, it suggests a lower severity.
Biothesiometer | The measurement will be taken during the baseline assessment and again after the completion of treatment.
  This objective measure is utilized to assess the vibratory pressure threshold in affected areas. It possesses the capability to detect various frequencies for vibratory pressure threshold assessment. It is regarded as a practical tool for evaluating both superficial and vibratory sensations. If there is an increased perception of frequency, it indicates that the vibratory pressure threshold is more severely affected.
NeuroQoL | The measurement will be taken during the baseline assessment and again after the completion of treatment.
  The Neuropathy-and Foot-Ulcer Specific Quality of Life Instrument is designed as a Likert scale and serves as a reliable method for assessing quality of life related to neuropathy. If the scoring indicates a higher value, it suggests that the disease is more severe.

SECONDARY OUTCOMES:
NPRS | The measurement will be taken during the baseline assessment and again after the completion of treatment.
  The Numeric Pain Rating Scale, ranging from 0 to 10, is employed as a subjective assessment tool to measure an individual's pain perception. In general, higher scores on the scale indicate a greater severity of pain linked to the disease.

CONTACTS AND LOCATIONS:
Overall Officials: Khushboo Kumari, BPT, (MPT), Principal Investigator — Maharishi Markandeshwar Instirtute of Physiotherapy and Rehabilitation, Ambala, Haryana, 133207
Locations (1):
- MMIPR, Ambāla, Haryana, India

IPD SHARING:
Plan to Share IPD: No